CLINICAL TRIAL: NCT02361073
Title: Event-related Potentials in Patients With Takotsubo Cardiomyopathy
Brief Title: The Role of Emotional Stress in Patients With Stress-induced Cardiomyopathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Magdeburg (Other)
Responsible Party: Principal Investigator, Dr. Samir Said, MD, University of Magdeburg
Other Study IDs: UM-PC-0813
Record Dates: First submitted 2013-01-09; First posted 2015-02-11 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-02

CONDITIONS: Takotsubo Cardiomyopathy
Keywords: Stress-induced cardiomyopathy; ERP
MeSH Terms: conditions — Takotsubo Cardiomyopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Takotsubo
- Healthy
- ACS

SUMMARY:
The event-related potentials may be different in patients with Takotsubo cardiomyopathy than in patients without Takotsubo.

DETAILED DESCRIPTION:
In patients with Takotsubo diagnosed by coronary angiography, the event-related potentials are investigated and compared with a control group, which consists of subjects without Takotsubo.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Written informed consent
* Takotsubo cardiomyopathy for group 1. ACS for group 3.

Exclusion Criteria:

* Psychiatric diseases
* Impaired versus, non compliant patients, heart disease for group 2.
* Takotsubo-like syndrome.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Takotsubo Cardiomyopathy compared with healthy subjects and patients with ACS.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2011-06; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Event-related potentials | up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Magdeburg, Magdeburg, Germany